CLINICAL TRIAL: NCT01927497
Title: Long-term Results of Biological Mesh Closure of the Pelvic Floor After Extralevator Abdominoperineal Resection for Rectal Cancer
Brief Title: Biological Mesh Closure of the Pelvic Floor After Extralevator Abdomino Perineal Resection for Rectal Cancer
Acronym: BIOPEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: LifeCell (Industry)
Responsible Party: Principal Investigator, P.J. Tanis, dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METC 2012_360; NTR3717 (Other: Nederlands Trial register)
Record Dates: First submitted 2013-08-19; First posted 2013-08-22 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Extralevator abdominoperineal resection; Biological Mesh; Primary closure
MeSH Terms: conditions — Rectal Neoplasms | interventions — strattice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biological mesh closure (Experimental): Biological mesh reconstruction of the pelvic floor after extralevator abdomino perineal resection
  Interventions: Procedure: Biological mesh assisted perineal closure
- Primary perineal closure (Active Comparator): Primary perineal closure after extralevator abdomino perineal resection
  Interventions: Procedure: Primary perineal closure

INTERVENTIONS:
Procedure: Biological mesh assisted perineal closure — The eAPR procedure will be performed in an identical way as described for the control arm of the study, and this is preferably followed by an omental plasty. The intervention in the experimental arm consists of suturing an acellular biological mesh derived from porcine dermis in the pelvic floor defect (Strattice™, 6x10 cm). The mesh will be sutured at each side of the coccyx or distal sacrum with Prolene or PDS to the discretion of the surgeon. Laterally, the mesh is attached to the remainings of the levator complex and, anteriorly, to the transverse perineal muscle or posterior vaginal wall. A suction drain will be inserted and positioned on top of the mesh. The perineal subcutaneous fat and skin will be subsequently closed in layers similar to primary simple closure as performed in the standard arm.
  Other Names: Biological Mesh; Strattice™; Strattice® Reconstructive Tissue Matrix; Lifecell; Porcine dermal Mesh
  Arms: Biological mesh closure
Procedure: Primary perineal closure — The perineal phase of the APR will be performed according to the principles of an extralevator APR, which means that the levator muscles will be laterally transected in order to leave a muscular cuff around the tumour. The coccyx will not be routinely resected, but only if indicated based on surgical exposure or oncological principles. The extent of excision of perineal skin and ischioanal fat will be as limited as oncologically justified. Preferably, an omental plasty is positioned in the pelvic cavity following resection. Closure of the perineum in the control arm consists of stitching the perineal subcutaneous fat together using interrupted Vicryl sutures in one or two layers. Subsequently, the skin will be closed using interrupted sutures according to the preference of the surgeon. Placement of a transabdominal or transperineal drain will be at the discretion of the surgeon.
  Other Names: Primary closure; Perineal wound closure
  Arms: Primary perineal closure

SUMMARY:
Rationale: Approximately 800 abdominoperineal resections (APR) are performed for rectal cancer each year in the Netherlands. The extralevator approach (eAPR) reduces the rate of positive margins and improves oncological outcome in distal rectal cancer. However, wider excisions increase wound healing problems and development of perineal hernia. This has resulted in a progressive increase of the use of musculocutaneous flaps and biological meshes associated with a substantial increase of costs, which is not supported by proper data.

Objective: The aim of this study is to determine the cost-effectiveness of pelvic floor reconstruction using a biological mesh after standardized eAPR with neo-adjuvant (chemo)radiotherapy.

Study design: This is a multicenter study in which patients undergoing an eAPR are randomized between standard care using primary closure of the perineum and the experimental arm with assisted closure using a biological mesh.

Study population: Patients with a clinical diagnosis of primary rectal cancer who are scheduled for eAPR after neo-adjuvant (chemo)radiotherapy. A total number of 104 patients will be randomized.

Intervention: The intervention in the experimental arm consists of suturing a biological mesh derived from porcine dermis in the pelvic floor defect, followed by perineal closure similar to the control arm.

Main study parameters/endpoints: The primary endpoint is the percentage of uncomplicated perineal wound healing (Souphampton wound score less than II at day 30). Secondary endpoints are hospital stay, incidence of perineal hernia, quality of life, and costs.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Both primary perineal closure and biological mesh assisted closure are being performed in daily clinical practise. The potential benefit resulting from participation of the study in patients randomized for biological mesh assisted closure may be a higher chance of uncomplicated perineal wound healing and lower perineal hernia rate. On the other hand, the use of a biological mesh has been associated with increased postoperative pain and seroma formation.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or higher.
2. Planned for eAPR for primary rectal cancer.
3. Life expectancy of more than 2 years.
4. Ability to return for all scheduled and required study visits.
5. Preoperative (chemo)radiotherapy.
6. Written informed consent for study participation.

Exclusion Criteria:

1. Previous pelvic irradiation for other cancers (i.e. prostate cancer).
2. Total exenteration or sacral resection above level S4/S5.
3. Sensitivity to porcine derived products or polysorbate.
4. Severe systemic diseases affecting wound healing (i.e. renal failure requiring dialysis, liver cirrhosis, and immune compromised status like HIV).
5. Collagen disorders (i.e. Marfan).
6. Enrolment in trials with overlapping primary endpoint or otherwise expected influence on wound healing (i.e. biological therapy like antiangiogenic agents).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-03-08 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2015-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gijsbert D. Musters, M.D., Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Willem A. Bemelman, Prof, PhD, M.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Harm J. Rutten, M.D. PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven; Baljit Singh, M.D. PhD, Principal Investigator — Leicester hospital, Leicester; Marcel G.W. Dijkgraaf, M.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Cener, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Musters GD, Bemelman WA, Bosker RJ, Burger JW, van Duijvendijk P, van Etten B, van Geloven AA, de Graaf EJ, Hoff C, de Korte N, Leijtens JW, Rutten HJ, Singh B, van de Ven A, Vuylsteke RJ, de Wilt JH, Dijkgraaf MG, Tanis PJ. Randomized controlled multicentre study comparing biological mesh closure of the pelvic floor with primary perineal wound closure after extralevator abdominoperineal resection for rectal cancer (BIOPEX-study). BMC Surg. 2014 Aug 27;14:58. doi: 10.1186/1471-2482-14-58. PMID 25163547

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biological Mesh Closure | Primary Perineal Closure
Started | 50 | 54
Completed | 48 | 53
Not Completed | 2 | 1
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: there were 2 drop-outs in the biological mesh group because no extralevator APR was performed, and 1 drop-out in the primary closure group because patient died preoperatively because of brain metastasis
Groups:
- Total: Total of all reporting groups
Arm/Group | Biological Mesh Closure | Primary Perineal Closure | Total
Number analyzed (Participants) | 48 | 53 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12) | 65 (12) | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 36 | 39 | 75

OUTCOME MEASURES:

1. Primary Outcome: 30-day Uncomplicated Perineal Wound Healing
Description: uncomplicated perineal wound healing is defined as a Souphampton wound score less than II
Time Frame: From operation to 30 days after the operation
Population: 2 drop-outs in the biological mesh group and 1 drop-out in de primary perineal closure group
Measure: Count of Participants; unit: Participants
Arm/Group | Biological Mesh Closure | Primary Perineal Closure
Number analyzed (Participants) | 48 | 53
Participants | 30 | 33

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Biological Mesh Closure | Primary Perineal Closure
All-Cause Mortality (participants affected / at risk) | 1/48 | 1/53
Serious Adverse Events (participants affected / at risk) | 20/48 | 20/53
Other Adverse Events (participants affected / at risk) | 20/48 | 20/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biological Mesh Closure (N=48) | Primary Perineal Closure (N=53)
surgical complication (Surgical and medical procedures) | 20 | 20 — Surgical complications are urinary retention, ileus, trocar hernia, postoperative bleeding, presacral fistula, stoma dysfunction, pneumonia, perineal hernia <90 days
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biological Mesh Closure (N=48) | Primary Perineal Closure (N=53)
surgical complication (Surgical and medical procedures) | 20 | 20 — Surgical complications are urinary retention, ileus, trocar hernia, postoperative bleeding, presacral fistula, stoma dysfunction, pneumonia, perineal hernia <90 days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes